CLINICAL TRIAL: NCT06123962
Title: Acute Lung/ Acute Respiratory Distress Syndrome and Extra-pulmonary Organ Injury Clinical Sub-phenotyping Study
Brief Title: ALI/ARDS Clinical Sub-phenotyping Study
Status: Recruiting | Type: Observational
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Jingen Xia, Clinical Professor, China-Japan Friendship Hospital
Other Study IDs: 2022YFC2504401
Record Dates: First submitted 2023-08-29; First posted 2023-11-09 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Acute Lung Injury/Acute Respiratory Distress Syndrome (ARDS)
Keywords: Acute Lung Injury/Acute Respiratory Distress Syndrome (ARDS); Sub-phenotypes; Treatment strategies
MeSH Terms: conditions — Acute Lung Injury; Respiratory Distress Syndrome | interventions — Bronchoalveolar Lavage Fluid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We plan to collect peripheral blood and bronchoalveolar lavage fluid.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Collect peripheral blood and bronchoalveolar lavage fluid — Peripheral venous blood will be collected and stored from the study participants at a total of five time points: Day 0, Day 1, Day 2, Day 3 after admission to the ICU, and the day of ICU discharge/death. The collection will be conducted after assessing the patients' eligibility for ARDS diagnosis. Each time point will involve the collection of one tube of peripheral venous blood, totaling 5 mL per sample.
  Within 24 hours after patients' admission to the ICU and meeting the assessment criteria for ARDS diagnosis, bronchoalveolar lavage fluid (BALF) will be collected and retained, totaling 10 mL.

SUMMARY:
1. Construct a structured clinical data and biosample information platform for Chinese patients with acute lung injury/ acute respiratory distress syndrome.
2. By deciphering the heterogeneity of patients with acute lung injury/ acute respiratory distress syndrome, achieve clinical, longitudinal physiological, and biological sub-phenotyping to guide individualized precision treatment and improve prognosis.

DETAILED DESCRIPTION:
Acute lung injury/ acute respiratory distress syndrome is one of the most common and complex critical illnesses in clinical practice, with a high mortality rate of 45% to 50%. Currently, effective therapeutic strategies for this condition are still lacking. Increasing evidence suggests that the significant heterogeneity of this disease plays a crucial role in the poor treatment outcomes and high mortality rates observed in patients. Therefore, this study aims to analyze the heterogeneity of acute lung injury/ acute respiratory distress syndrome patients and establish a clinical classification system for acute lung and extrapulmonary organ injuries.

The objectives of this study include establishing a nationwide clinical database and biobank for acute lung injury / acute respiratory distress syndrome by collecting clinical data and biological samples from various provinces. By overcoming the barriers posed by diverse and heterogeneous data sources, mathematical and machine learning models will be utilized to construct clinical, physiological, and biological classification systems for acute lung and extrapulmonary organ injuries. The proposed classification model will be validated multiple times using international public databases and prospective acute lung injury/acute respiratory distress syndrome cohorts to ensure its stability and generalizability. The mapping relationship between different classifications and patient prognosis as well as treatment responsiveness will be explored.

Moreover, a machine learning-based supervised technique will be applied to develop a bedside simplified model (Point-of-Care model) and establish a bedside clinical classification decision system. Ultimately, this research aims to provide a foundation for standardized and precision-guided clinical diagnostic and therapeutic pathways, promoting improved treatment outcomes and overall prognosis in acute lung injury/ acute respiratory distress syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria for Acute Respiratory Distress Syndrome (ARDS) according to the updated global definition in 2023.
* The patient or their legal representative signs an informed consent form.

Exclusion Criteria:

* Individuals aged less than 18 years old.
* Those who refuse to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Updated global diagnostic criteria for Acute Respiratory Distress Syndrome (ARDS) in 2023 are as follows:
  Supportive respiratory criteria: Endotracheal intubation, or non-invasive ventilation (NIV)/continuous positive airway pressure (CPAP) with minimum expiratory positive airway pressure (EPAP) ≥ 5 cmH2O, or high-flow nasal oxygen therapy with a minimum flow rate ≥ 30 L/min.
  Hypoxemia criteria: Arterial partial pressure of oxygen to fraction of inspired oxygen ratio (PaO2/FiO2) ≤ 300 mmHg, or peripheral oxygen saturation to fraction of inspired oxygen ratio (SpO2/FiO2) ≤ 315 mmHg, with simultaneous peripheral oxygen saturation (SpO2) ≤ 97%.
  Radiographic criteria: Chest X-ray, chest computed tomography (CT), or trained ultrasound confirming bilateral pulmonary opacities.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2023-12-14 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
ICU mortality | up to 12 weeks
  In ICU mortality
hospital mortality | up to 24 weeks
  In hospital mortality

SECONDARY OUTCOMES:
28 days without mechanical ventilation | up to 28 days
  28 days without mechanical ventilation
length of stay in the ICU | up to 12 weeks
  length of stay in the ICU
Total length of hospital stay | up to 24 weeks
  Total length of hospital stay
Mortality at 1 year after discharge | through study completion, an average of 1 year
  Mortality at 1 year after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Jingen Xia, Study Director — China-Japan Friendship Hospital
Locations (1):
- Jingen Xia, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thompson BT, Chambers RC, Liu KD. Acute Respiratory Distress Syndrome. N Engl J Med. 2017 Aug 10;377(6):562-572. doi: 10.1056/NEJMra1608077. No abstract available. PMID 28792873
- [Background] Huang X, Zhang R, Fan G, Wu D, Lu H, Wang D, Deng W, Sun T, Xing L, Liu S, Wang S, Cai Y, Tian Y, Zhang Y, Xia J, Zhan Q; CHARDSnet group. Incidence and outcomes of acute respiratory distress syndrome in intensive care units of mainland China: a multicentre prospective longitudinal study. Crit Care. 2020 Aug 20;24(1):515. doi: 10.1186/s13054-020-03112-0. PMID 32819400
- [Background] Reilly JP, Calfee CS, Christie JD. Acute Respiratory Distress Syndrome Phenotypes. Semin Respir Crit Care Med. 2019 Feb;40(1):19-30. doi: 10.1055/s-0039-1684049. Epub 2019 May 6. PMID 31060085
- [Background] Shah FA, Meyer NJ, Angus DC, Awdish R, Azoulay E, Calfee CS, Clermont G, Gordon AC, Kwizera A, Leligdowicz A, Marshall JC, Mikacenic C, Sinha P, Venkatesh B, Wong HR, Zampieri FG, Yende S. A Research Agenda for Precision Medicine in Sepsis and Acute Respiratory Distress Syndrome: An Official American Thoracic Society Research Statement. Am J Respir Crit Care Med. 2021 Oct 15;204(8):891-901. doi: 10.1164/rccm.202108-1908ST. PMID 34652268
- [Background] Calfee CS, Delucchi K, Parsons PE, Thompson BT, Ware LB, Matthay MA; NHLBI ARDS Network. Subphenotypes in acute respiratory distress syndrome: latent class analysis of data from two randomised controlled trials. Lancet Respir Med. 2014 Aug;2(8):611-20. doi: 10.1016/S2213-2600(14)70097-9. Epub 2014 May 19. PMID 24853585